CLINICAL TRIAL: NCT04385940
Title: Improving Vitamin D Status in the Management of COVID-19
Brief Title: Vitamin D and COVID-19 Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00100606
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose vitamin D (Experimental): Ddrops® products,Vitamin D3, 50,000 IU, Oral
  Interventions: Dietary Supplement: Ddrops® products, 50,000 IU, Oral
- Low dose vitamin D (Active Comparator): Vitamin D3 1000IU
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Ddrops® products, 50,000 IU, Oral — Vitamin D3
  Arms: High dose vitamin D
Dietary Supplement: Vitamin D3 — Vitamin D3 1000IU
  Arms: Low dose vitamin D

SUMMARY:
A novel coronavirus disease 2019 (COVID-19) outbreak is a global dramatic pandemic that is immeasurably impacting the communities. Due to lack of data, symptomatic management is used for COVID-19 infection including oxygen therapy and mechanical ventilation for those with severe infection. Considering immunomodulatory, anti-inflammatory anti-fibrotic and anti-oxidant actions of vitamin D, it's safety and ease of administration, as well as direct effects of vitamin D on immune cell proliferation and activity, pulmonary ACE2 expression and reducing surface tension, evaluation of vitamin D supplementation as an adjuvant therapeutic intervention could be of substantial clinical and economic significance. High prevalence of vitamin D deficiency in elderly, smokers, patients with chronic diseases and excess uptake by adipose tissue in obesity make investigations of its role as a secondary therapeutic agent in COVID-19 conceivable. It should be necessary to monitor serum 25(OH)D levels in all inpatient and outpatient populations with COVID-19 to identify the importance of maintaining or promptly increasing circulating levels of 25(OH)D into the optimal range of 100-150 nmol/L.

The aim of this study is to conduct a double blind, randomized, controlled three weeks clinical trial on the efficacy of vitamin D (daily low dose versus weekly high dose) in COVID-19 patients in order to determine the relationship between baseline vitamin D deficiency and clinical characteristics and to asses patients' response to vitamin D supplementation in week three and determine its association with disease progression and recovery.

Subjects who are randomized to high-dose will be asked to take 50,000 IU for two times during the first week and one dose over second and third weeks to quickly raise their serum levels. Subjects in the low-dose arm will take vitamin D 1000 IU daily for three weeks.

DETAILED DESCRIPTION:
In-patients

1. Determine the frequency of low serum Vit D levels (<50 nmol/L) in COVID-19 patients.
2. Determine the relationship between baseline vitamin D status and disease severity, laboratory biochemical tests of white blood cell count (WBC), C-reactive protein (CRP), lymphocyte count, leukocytes counts and neutrophil-lymphocyte-ratio (NLR), lactate dehydrogenase, IL-6, IL-1beta, TNF-alpha platelet count, albumin, and serum ferritin, required hospitalization and intensive care unit (ICU) admission.
3. Asses patients' initial response to vitamin D supplementation in week one and determine its association with disease progression and recovery.
4. Compare disease severity and progression, laboratory biochemical tests of white blood cell count (WBC), C-reactive protein (CRP), lymphocyte count, lactate dehydrogenase, IL-6, IL-1beta, TNF-alpha, platelet count, albumin, and serum ferritin, hospital admission and length of stay, duration of mechanical ventilation, hospital mortality and respiratory failure differ between the early responder and non-responder groups.

Out-patients

1. Determine the frequency of low serum Vit D levels (<50 nmol/L) in COVID-19 patients.
2. Determine the relationship between baseline vitamin D deficiency and clinical characteristics.
3. Asses patients' response to vitamin D supplementation in week three and determine its association with disease progression and recovery

ELIGIBILITY:
Inclusion Criteria:

Patients with COVID-19:

* ≥ 17 years old
* Both sexes

Exclusion Criteria:

* Patients with dementia, learning disability, mental health needs and alcohol or drug dependency, pregnant women will be excluded.
* Patients with sarcoidosis, hypercalcemia, known vitamin D intolerance

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Symptoms recovery | Time from onset of intervention to day 21
  Number of Participants whose symptoms recovered over three weeks

SECONDARY OUTCOMES:
Hospitalization | Between diagnosis and day 21
  Number of patients who required hospitalization
Blood white blood cell count (WBC) | At day 0 before starting intervention and day 21 of intervention
  x 109/L
Duration of mechanical ventilation | Between diagnosis and day 21
  If patients required mechanical ventilation at any time after diagnosis
Duration of hospitalization | Between diagnosis and day 21
  Length of stay in hospital (days)
Intensive care unit (ICU) admission | Between diagnosis and day 21
  Number of patients who required ICU
Duration of ICU stay | Between diagnosis and day 21
  Length of stay in ICU
Blood C-reactive protein (CRP) | Baseline and day 21
  mg/L
Blood Lymphocyte count | Baseline and day 21
  number of lymphocytes in 1 microliter (µL) of blood
Blood Ferritin | Baseline and day 21
  ng/mL
Blood platelet count | Baseline and day 21
  platelets per microliter of blood
Blood interleukin-6 (IL-6) | Baseline and day 21
  pg/mL
Blood Tumor Necrosis Factor alpha (TNF) | Baseline and day 21
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Montano-Loza, MD, MSc, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided